CLINICAL TRIAL: NCT06842368
Title: Immediate Implant Placement Using Xenograft As Space Filling Material Mixed with Vitamin D Versus Hyaluronic Acid in Posterior Mandible Region: a Randomized Controlled Clinical Trial.
Brief Title: Immediate Implant Placement Using Xenograft Mixed with Vitamin D Versus Hyaluronic Acid.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ammar Mohamad Adib Eiz Eddin, Master's degree candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A.M.A.E
Record Dates: First submitted 2025-02-03; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Immediate Implant Placement
Keywords: Hyaluronic acid; Vitamin D; Xenograft; Immediate Implant
MeSH Terms: interventions — Hyaluronic Acid; Vitamin D

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial. Parallel group study. Allocation Ratio 1:1.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Each patient will be given a code by the researcher and the observers will be blind to which group this case belong. Patients, radiographic outcome assessor and statistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D mixed with Xenograft as space filling material after placement of immediate implant. (Experimental): Careful extraction of the selected tooth will initiated using sharp periotome to sever the periodontal ligament attachments while preserving the surrounding alveolar bone and interdental papilla and followed by using extraction forceps. Meticulous mechanical debridement of the extraction socket will be carried out using bone curette to remove any soft tissue remnants or granulation tissue. All debris will washed out using copious saline irrigation. Implant osteotomy will then initiated engaging the furcation of the alveolus along with the remaining apical bone and while maintain jumping gap more than 2 mm between the implant platform and the alveolar. the jumping space will packed using Xenograft with particle size ranging from 0.25 to 1 mm and it will be mixed with Vitamin D and the socket will sealed using 4-0 resorbable sutures.
  Interventions: Procedure: Vitamin D
- Hyaluronic acid mixed with Xenograft as space filling material after placement of immediate implant. (Active Comparator): Careful extraction of the selected tooth will initiated using sharp periotome to sever the periodontal ligament attachments while preserving the surrounding alveolar bone and interdental papilla and followed by using extraction forceps. Meticulous mechanical debridement of the extraction socket will be carried out using bone curette to remove any soft tissue remnants or granulation tissue. All debris will washed out using copious saline irrigation. Implant osteotomy will then initiated engaging the furcation of the alveolus along with the remaining apical bone and while maintain jumping gap more than 2 mm between the implant platform and the alveolar. the jumping space will packed using Xenograft with particle size ranging from 0.25 to 1 mm and it will be mixed with hyaluronic acid and the socket will sealed using 4-0 resorbable sutures.
  Interventions: Procedure: Hyaluronic Acid (HA)

INTERVENTIONS:
Procedure: Hyaluronic Acid (HA) — Hyaluronic acid is one of the essential components of extracellular matrix, which plays a predominant role in tissue morphogenesis, cell migration, differentiation, and adhesion. It has been recently reported that hyaluronic acid increases osteoblastic bone formation in vitro through increased mesenchymal cell differentiation and migration.
  It has demonstrated that Hyaluronic acid not only acted as a carrier of growth factors and cell but also stimulated bone formation through chemotaxis, proliferation and differentiation of mesenchymal cells into osteoblasts.
  Although Hyaluronic acid shares bone induction properties with growth factors as bone morphogenic protein 2 and osteopontin
  Arms: Hyaluronic acid mixed with Xenograft as space filling material after placement of immediate implant.
Procedure: Vitamin D — It was shown that locally applied vitamin D3 in combination with bovine bone mineral matrix improved the bone formation and strengthened the site of the fracture in ovariectomized rats.
  Local application of vitamin D3 also proved to be promising in promoting osteo- genesis and mineralization for restoration of bone defects. Grounding on this incites, it has been suggested that vitamin D3 might exert a positive local effect on alveolar bone regeneration
  Arms: Vitamin D mixed with Xenograft as space filling material after placement of immediate implant.

SUMMARY:
Immediate implant placement using xenograft as space filling material mixed with vitamin D versus hyaluronic acid in posterior mandible region This study aims to evaluate implant stability and density after placement of immediate implant and Xenograft mixed with Hyaluronic acid or Vitamin D at posterior mandible region

DETAILED DESCRIPTION:
Dental implants in fresh extraction sockets and healed sites have a erratic morphology, creating a wide space defect between the implant and buccal alveolar bone. This defect is critical for implant success, known as a jumping gap. Proper management of this space is essential for esthetic and functional success. Studies show adequate bone fill can be achieved in jumping gaps, but wider gaps increase implant body exposure risk.

The application of biological mediators embedded in the biomaterial can induce specific cell and tissue response, which can improve bone quality and quantity. Dental research has focused on improving bone substitutes by morphologic or bio- chemical modification.

ELIGIBILITY:
Inclusion Criteria:

Age: 18-60.

* Systemically healthy patients indicated for single or multiple immediate implants in posterior teeth region.
* Absence of any peri-apical pathosis.
* Patients with intact buccal plate of bone.
* Patients with adequate bone volume for the dental implant procedure.
* Patient with good oral hygrine

Exclusion Criteria:

* Heavy Smokers.
* Systemic disease that may affect the final outcome of the surgical procedure.
* No or poor patient's compliance.
* Patients with psychological problems.
* Pathology at the site of intervention.
* Patient with vit d deficiency

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Implant secondary stability | after 6 months
  To evaluate the implant stability by Any-check device.

SECONDARY OUTCOMES:
Density of bone around implant | after 6 months
  Cone beam computed tomography CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry ,Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abd Elwahap, Mohammad et al. "Effect of Xenograft Alone versus Xenograft Mixed with Vitamin-D On Preservation of Alveolar Sockets of Chronically Infected Teeth." Al-Azhar Journal of Dental Science (2024): n. pag.
- [Background] ⦁ Elgazzar, A., Yousef, E., Amer, M. Effect of Hyaluronic Acid Mixed with Biphasic Calcium Phosphate on Bone Healing Around Immediately Placed Implants in the Posterior Area of the Mandible. Egyptian Dental Journal, 2023; 69(4): 2631-2641. doi: 10.21608/edj.2023.227200.2669